CLINICAL TRIAL: NCT00367432
Title: A Multicenter, Open, Long-term Follow-up Study to Evaluate the Safety and Efficacy of L059 (Levetiracetam) at Individual Optimal Dose Ranging From 500 to 3000 mg/Day in Twice Daily Administration in Subjects From 16 to 65 Years With Epilepsy Suffering From Partial Onset Seizures Whether or Not Secondarily Generalized Who Completed in a Previous Study
Brief Title: A Long Term Follow up Administration Study of L059 (Levetiracetam) in Epilepsy Patients With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01222; 2014-004334-26 (EudraCT Number)
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2015-04

CONDITIONS: Epilepsies; Partial
Keywords: Epilepsies; Partial; Keppra; levetiracetam
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental): Levetiracetam 500 mg/day to 3000 mg/day , tablets twice daily (morning and evening orally) during the study period (until the time of approval granted).
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam 500 mg/day to 3000 mg/day , tablets twice daily (morning and evening orally) during the study period (until the time of approval granted).
  Other Names: Keppra

SUMMARY:
This study is planned to evaluate the safety and efficacy of L059 (levetiracetam) in long-term administration in patients who completed N01020 [NCT00160165] or N01221 [NCT00280696].

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in study N01221 [NCT00280696] and completed the evaluation period and transition period or patients who participated in study N01020 [NCT00160615]

Exclusion Criteria:

* Female patients during pregnancy, delivery and lactation, or suspected of pregnancy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2006-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (53):
- Japan (53):
  - Aichi-gun, Aichi-ken
  - Nagoya, Aichi-ken
  - Hirosaki, Aomori
  - Matsudo, Chiba
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kurume, Fukuoka
  - Fukuyama, Hiroshima
  - Asahikawa, Hokkaido
  - Hakodate, Hokkaido
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Kahoku-gun, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Zentsujichó, Kagawa-ken
  - Kōshi, Kumamoto
  - Tsu, Mie-ken
  - Iwanuma, Miyagi
  - Sendai, Miyagi
  - Ōmura, Nagasaki
  - Kashihara, Nara
  - Nagaoka, Niigata
  - Beppu, Oita Prefecture
  - Izumi, Osaka
  - Neyagawa, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Iruma-gun, Saitama
  - Shimotsuga-gun, Tochigi
  - Shimotsuke, Tochigi
  - Komatsushimachō, Tokushima
  - Chiyoda-Ku, Tokyo
  - Kodaira, Tokyo
  - Kokubunji, Tokyo
  - Shinjuku-ku, Tokyo
  - Taito-ku, Tokyo
  - Ube, Yamaguchi
  - Aomori
  - Chiba
  - Fukuoka
  - Fukushima
  - Gifu
  - Hiroshima
  - Kagoshima
  - Kumamoto
  - Kyoto
  - Miyazaki
  - Niigata
  - Okayama
  - Osaka
  - Shizuoka
  - Toyama
  - Yamagata

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Full Analysis Set (FAS) includes all subjects to whom the investigational products are assigned after registration, excluding those with serious Good Clinical Practice violations , subjects not administered the investigational products and subjects for whom no data is available after assignment of the investigational products.
Pre-assignment Details: Eligible subjects from preceding study N01221 [NCT00280696] entered the First Period of this study and those subjects from N01221 [NCT00280696] who completed the First Period and subjects from the study N01020 [NCT00160615] entered the Second Period.
  Participant Flow and Baseline Characteristics refer to the FAS.
Groups:
- Levetiracetam N01221 [NCT00280696]: N01221 [NCT00280696] was a double-blind, randomized, multicenter, placebo controlled 5 parallel groups, confirmatory trial to evaluate the efficacy and safety of Levetiracetam.
- Levetiracetam N01020 [NCT00160615]: N01020 [NCT00160615] was an open-label follow-up study to evaluate safety and efficacy of Levetiracetam.
Period: First Period (16 Weeks)
Arm/Group | Levetiracetam N01221 [NCT00280696] | Levetiracetam N01020 [NCT00160615]
Started | 313 (Eligible subjects from preceding study N01221 [NCT00280696] entered the First Period of N01222) | 0
Completed | 275 | 0
Not Completed | 38 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Lack of Efficacy | 24 | 0
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Other Reason | 2 | 0
Period: Second Period (up to 54 Months)
Arm/Group | Levetiracetam N01221 [NCT00280696] | Levetiracetam N01020 [NCT00160615]
Started | 275 (275 subjects from N01221 [NCT00280696] completed First Period and entered Second Period of N01222) | 85 (85 subjects from N01020 [NCT00160615] entered Second Period of N01222)
Completed | 188 | 69
Not Completed | 87 | 16
Not completed — Adverse Event | 14 | 3
Not completed — Lack of Efficacy | 59 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Other Reason | 6 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam
Number analyzed (Participants) | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.68 (11.18)
Age, Customized [Number; unit: participants]
  Between 16 and 65 years | 398
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 202
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 396
  Asian (other than Japanese) | 2
Region of Enrollment [Number; unit: participants]
  Japan | 398
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 60.39 (13.64)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Treatment-emergent Adverse Events During the Study Period (Until the Time of Approval Granted)
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with the pharmaceutical product.
  Occurrence of treatment-emergent AEs is reported by the number of subjects with at least one treatment-emergent AE.
Time Frame: During the study period from Visit 1 (Week 0) to the Follow-up Visit (up to Month 60) until the time of approval granted
Population: Safety Set includes all subjects from N01221 [NCT00280696] and N01020 [NCT00160615] administered the investigational products at least once.
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 398
participants | 381

2. Secondary Outcome: Change From Baseline in N01221 [NCT00280696] in Partial (Type 1) Seizure Frequency Per Week During the First 16-week Period in This Study
Description: The change in partial (type 1) seizure frequency from Baseline is given as a percent reduction computed as:
  [ Weekly partial seizure frequency (Baseline)- Weekly partial seizure frequency (Evaluation Period)]/ [Weekly partial seizure frequency (Baseline)] x 100.
  Positive values in percent reduction means that the value has decreased from Baseline during the first 16-week Period.
  Partial (Type I) seizures can be classified into one of the following three groups: Simple partial seizures, Complex partial seizures, Partial seizures evolving to secondarily generalized seizures.
Time Frame: Baseline in N01221 [NCT00280696], the First 16-week Evaluation Period from Visit 1 (Week 0) to Visit 5 (Week 16) in this study
Population: Full Analysis Set (FAS).
Measure: Median (Inter-Quartile Range); unit: Percent Reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 313
Percent Reduction | 22.00 (53.04) [-11.00 to 46.71]

3. Secondary Outcome: Seizure Frequency Per Week in Partial Seizures During the First 16-week Period in This Study
Description: Partial (Type I) seizures can be classified into one of the following three groups: Simple partial seizures, Complex partial seizures, Partial seizures evolving to secondarily generalized seizures.
Time Frame: First 16-week Evaluation Period from Visit 1 (Week 0) to Visit 5 ( Week 16)
Population: Full Analysis Set (FAS).
Measure: Median (Inter-Quartile Range); unit: Seizures Per Week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 313
Seizures Per Week | 2.13 (7.32) [1.06 to 5.23]

4. Secondary Outcome: Response Status (Patients With a Percent Reduction in Partial Seizure Frequency of at Least 50% During the First 16-week Period in This Study From Baseline in N01221)
Description: The percent reduction from Baseline was computed as:
  [ Weekly seizure frequency (Baseline)- Weekly seizure frequency (Evaluation Period)]/ [Weekly seizure frequency (Baseline)] x 100.
  Responders are those patients with a percent reduction in partial seizure frequency of at least 50% from Baseline to first Evaluation Period in partial seizure frequency per week.
  Partial (Type I) seizures can be classified into one of the following three groups: Simple partial seizures, Complex partial seizures, Partial seizures evolving to secondarily generalized seizures.
Time Frame: as for outcome 2
Population: Full Analysis Set (FAS).
Measure: Number; unit: Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 313
Participants
  Responders | 74
  Non-responders | 239

5. Secondary Outcome: Change From Baseline in N01221 [NCT00280696] in Simple Partial Seizure Frequency Per Week During the First 16-week Period in This Study
Description: Change in simple partial seizure frequency is given as a percent reduction computed as:
  [ Weekly simple partial seizure frequency (Baseline)- Weekly simple partial seizure frequency (Evaluation Period)]/ [Weekly simple partial seizure frequency (Baseline)] x 100.
  Positive values in percent reduction means that the value has decreased from Baseline during the first 16-week Period.
  Partial (Type I) seizures can be classified into one of the following three groups: Simple partial seizures, Complex partial seizures, Partial seizures evolving to secondarily generalized seizures.
Time Frame: as for outcome 2
Population: Subset of the FAS population excluding subjects with seizure counts equal to zero during Baseline and Evaluation Period for Simple Partial Seizures.
Measure: Median (Inter-Quartile Range); unit: Percent Reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 173
Percent Reduction | 39.84 (139.32) [-17.19 to 94.96]

6. Secondary Outcome: Change From Baseline in N01221 [NCT00280696] in Complex Partial Seizure Frequency Per Week During the First 16-week Period in This Study
Description: Change in complex partial seizure frequency is given as a percent reduction computed as:
  [ Weekly complex partial seizure frequency (Baseline)- Weekly complex partial seizure frequency (Evaluation Period)]/ [Weekly complex partial seizure frequency (Baseline)] x 100.
  Positive values in percent reduction means that the value has decreased from Baseline during the first 16-week Period.
  Partial (Type I) seizures can be classified into one of the following three groups: Simple partial seizures, Complex partial seizures, Partial seizures evolving to secondarily generalized seizures.
Time Frame: as for outcome 2
Population: Subset of the FAS population excluding subjects with seizure counts equal to zero during Baseline and Evaluation Period for Complex Partial Seizures.
Measure: Median (Inter-Quartile Range); unit: Percent Reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 285
Percent Reduction | 20.59 (85.94) [-15.24 to 52.94]

7. Secondary Outcome: Change From Baseline in N01221 [NCT00280696] in Secondary Generalized Seizure Frequency Per Week During the First 16-week Period in This Study
Description: Change in secondary generalized seizure frequency is given as a percent reduction computed as:
  [ Weekly sec. generalized seizure frequency (Baseline)- Weekly sec. generalized seizure frequency (Evaluation Period)]/ [Weekly sec. generalized seizure frequency (Baseline)] x 100.
  Positive values in reduction means the value decreased from Baseline during the first 16-week Period.
  Secondary generalized seizures belong to one of the 3 groups:
  * Simple partial sz evolving to gen sz
  * Complex partial sz evolving to gen sz
  * Simple partial sz evolving to Complex partial sz evolving to gen sz
Time Frame: as for outcome 2
Population: Subset of the FAS population excluding subjects with seizure counts equal to zero during Baseline and Evaluation Period for Secondary Generalized Seizures.
Measure: Median (Inter-Quartile Range); unit: Percent Reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 87
Percent Reduction | 76.56 (249.71) [23.11 to 100.00]

8. Secondary Outcome: Change From Baseline in N01221 [NCT00280696] in Simple and Complex Partial Seizure Frequency Per Week During the First 16-week Period in This Study
Description: Change in simple and complex partial seizure frequency is given as a percent reduction computed as (simple and complex partial seizure frequency := A):
  [ Weekly A (Baseline)- Weekly A (Evaluation Period)]/ [Weekly A (Baseline)] x 100.
  Positive values in percent reduction means that the value has decreased from Baseline during the first 16-week Period.
  Partial (Type I) seizures can be classified into one of the following three groups: Simple partial seizures, Complex partial seizures, Partial seizures evolving to secondarily generalized seizures.
Time Frame: as for outcome 2
Population: Subset of the FAS population excluding subjects with seizure counts equal to zero during Baseline and Evaluation Period for Simple and Complex Partial Seizures.
Measure: Median (Inter-Quartile Range); unit: Percent Reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 308
Percent Reduction | 20.71 (63.01) [-13.17 to 47.42]

9. Secondary Outcome: Change From Baseline in N01221 [NCT00280696] in Other Types of Seizure Frequency Per Week During the First 16-week Period in This Study
Description: Change in other types of seizure frequency is given as a percent reduction computed as (other types of seizure frequency:= B):
  [ Weekly B (Baseline)- Weekly B (Evaluation Period)]/ [Weekly B (Baseline)] x 100.
  Positive values in percent reduction means that the value has decreased from Baseline during the first 16-week Period.
  Other types of Seizures are all seizures except Partial Seizures (Type 1).
Time Frame: as for outcome 2
Population: Subset of the FAS population excluding subjects with seizure counts equal to zero during Baseline and Evaluation Period for Other Types of Seizures.
Measure: Median (Inter-Quartile Range); unit: Percent Reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 5
Percent Reduction | 66.47 (71.28) [7.48 to 100.00]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 60 months from Visit 1 (Week 0) over the First and Second Period until Down-titration and Follow up.
Description: Adverse Events refer to the Safety Set (SS). SS includes all subjects from studies N01221 [NCT00280696] and N01020 [NCT00160615] administered the investigational products at least once.
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 64/398
Other Adverse Events (participants affected / at risk) | 369/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=398)
Abortion Complete (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abortion Induced (Surgical and medical procedures) | 2 (2)
Acute Psychosis (Psychiatric disorders) | 1 (1)
Acute Sinusitis (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Anticonvulsant Drug Level Increased (Investigations) | 2 (2)
Anticonvulsant Toxicity (Injury, poisoning and procedural complications) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Brain Operation (Surgical and medical procedures) | 1 (1)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Complex Partial Seizures (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Drug Withdrawal Convulsions (Nervous system disorders) | 1 (1)
Electrocardiogram ST Segment Elevation (Investigations) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 5 (5)
Eyelid Ptosis (Eye disorders) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroenteritis Escherichia Coli (Infections and infestations) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Head Titubation (Nervous system disorders) | 1 (1)
Ideas of Reference (Psychiatric disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infected Epidermal Cyst (Infections and infestations) | 1 (1)
Injection Site Infection (Infections and infestations) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1)
Jaw Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Lactation Disorder (Reproductive system and breast disorders) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Medical Diet (Surgical and medical procedures) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental Disorder (Psychiatric disorders) | 1 (1)
Morose (Psychiatric disorders) | 1 (3)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia Mycoplasmal (Infections and infestations) | 1 (1)
Postictal State (Nervous system disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Rectal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 3 (3)
Skull Fracture (Injury, poisoning and procedural complications) | 1 (1)
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Status Epilepticus (Nervous system disorders) | 5 (9)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Sudden Unexplained Death in Epilepsy (General disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Urethral Stenosis (Renal and urinary disorders) | 1 (2)
Wisdom Teeth Removal (Surgical and medical procedures) | 1 (1)
Colonic Polyp (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=398)
Abdominal Pain (Gastrointestinal disorders) | 38 (67)
Abdominal Pain Upper (Gastrointestinal disorders) | 20 (40)
Constipation (Gastrointestinal disorders) | 45 (70)
Diarrhoea (Gastrointestinal disorders) | 69 (128)
Nausea (Gastrointestinal disorders) | 44 (53)
Stomatitis (Gastrointestinal disorders) | 42 (75)
Toothache (Gastrointestinal disorders) | 21 (32)
Vomiting (Gastrointestinal disorders) | 40 (85)
Pyrexia (General disorders) | 52 (95)
Seasonal Allergy (Immune system disorders) | 29 (43)
Dental Caries (Infections and infestations) | 42 (49)
Gastroenteritis (Infections and infestations) | 27 (34)
Influenza (Infections and infestations) | 32 (32)
Nasopharyngitis (Infections and infestations) | 308 (1360)
Pharyngitis (Infections and infestations) | 25 (38)
Rhinitis (Infections and infestations) | 22 (26)
Contusion (Injury, poisoning and procedural complications) | 110 (237)
Excoriation (Injury, poisoning and procedural complications) | 52 (85)
Injury (Injury, poisoning and procedural complications) | 33 (39)
Joint Sprain (Injury, poisoning and procedural complications) | 27 (37)
Laceration (Injury, poisoning and procedural complications) | 20 (23)
Skin Laceration (Injury, poisoning and procedural complications) | 31 (53)
Thermal Burn (Injury, poisoning and procedural complications) | 36 (43)
Weight Decreased (Investigations) | 28 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (34)
Back Pain (Musculoskeletal and connective tissue disorders) | 45 (70)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (27)
Dizziness (Nervous system disorders) | 63 (92)
Epilepsy (Nervous system disorders) | 31 (37)
Headache (Nervous system disorders) | 96 (261)
Somnolence (Nervous system disorders) | 159 (226)
Insomnia (Psychiatric disorders) | 24 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (25)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 32 (60)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 20 (26)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 33 (46)
Eczema (Skin and subcutaneous tissue disorders) | 47 (61)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (25)
Rash (Skin and subcutaneous tissue disorders) | 26 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days